CLINICAL TRIAL: NCT04102787
Title: The Effect of Cardiac Educational Program on Level of Knowledge and Satisfaction Among Coronary Artery Disease Patients in North of Jordan
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jordan University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB in KAUH#
Record Dates: First submitted 2019-05-12; First posted 2019-09-25 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Coronary Artery Disease
Keywords: coronary artery disease, educational program, patient satisfaction, patient knowledge.
MeSH Terms: conditions — Coronary Artery Disease; Patient Satisfaction

STUDY DESIGN:
Intervention Model Description: pre and post true experimental with two groups control and experimental
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): Experimental group who received the Cardiac educational program and will be applied for Coronary Artery Disease patients, and measure the level of knowledge and satisfaction in pre and post test.
  Interventions: Other: cardiac educational program
- control group (No Intervention): Control group who received the usual care and measure the level of knowledge and satisfaction in pre and post test.

INTERVENTIONS:
Other: cardiac educational program — "Love your Heart" is a Heart Foundation program (2016), the Arabic version will be used as the educational program in this study. The programme has been adopted from relevant articles in the evidence- based literature. The program is a guide to support recovery and good heart health. It includes the following: anatomy and physiology of the heart, causes, symptoms and risk factors of CAD, healthy diet, physical activity, weight management, and risk factors management.
  Arms: experimental group

SUMMARY:
Background: Although patients' education programs improve health-related knowledge that promote individual capacity to understand basic health information, there is a scarcity in the studies that address cardiac educational programs for patients with coronary artery diseases in Jordan and their impact on patients' health outcomes.

Aim: the aims of this study are to assess the level of knowledge and satisfaction of patients with coronary artery disease and to evaluate the effect of implementing a cardiac educational program on patient's level of knowledge and satisfaction.

Methods: This study will be carried out using a true experimental two groups pre and post- test. The necessary information will be collected from 138 patients with CAD in the north of Jordan using the Coronary Artery Disease Education Questionnaire (CADE-Q) and the Patient Satisfaction Scale (PSS).

The expected outcomes include establishing foundational knowledge about the effectiveness of cardiac educational program on patient health related out comes. Evidence on the effect of cardiac educational program will help patients to recover from a heart attacks, prevent future heart problems, hospital stays and death related to heart problems as well as making a necessary life style changes.

Keywords: coronary artery disease, educational program, patient satisfaction, patient knowledge.

ELIGIBILITY:
Inclusion Criteria:

1. mentally competent since cognitive impairment negatively affects the comprehension of the cardiac educational program content
2. able to communicate verbally
3. able to read and write Arabic language
4. more than 18 years
5. stable and the previous attack not less than 24 hours

Exclusion Criteria:

* Exclusion criterion included patients with life- threatening comorbidities like (heart failure (HF), Valve Diseases, Chronic Obstructive Pulmonary Disease (COPD), patients with Pacemaker or Implanted Cardioverter Defibrillator (ICD), and any type of chronic cardiac arrythmias.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2018-10-28 (Actual); Primary Completion 2018-10-28 (Actual); Study Completion 2020-12-11 (Estimated)

PRIMARY OUTCOMES:
level of knowledge | up to one month
  level of knowledge using The Coronary Artery Disease Education Questionnaire Short Version (CADE- Q SV) . The CADEQ-SV was designed to be a true/false/I do not know questionnaire, with 20 items (4 in each domain). The CADE- Q SV was divided into four subscales. These include the following: firstly, items number 1, 3, 6,11 and 15 are related to the first part which covers the medical condition. Secondly, items number 2, 12, 16, and 18 are related to the second part which covers the risk factors. Thirdly, items number 5,9,14, and 20 deal with the third part which covers the nutrition. Fourthly, items number 4, 18, 13, and 17 deal with the fourth part which covers the physical exercise. Finally, items number 7, 10, and 19 are concerned with the fourth part which covers the psychological factors. Each correct answer equals
  1 point; therefore, the maximum score possible is 20 overall

SECONDARY OUTCOMES:
Patient satisfaction | up to one month
  Patient Satisfaction Scale (PSS) to measure the satisfaction level in likert scale (strongly disagree, disagree, not sure agree, and strongly agree).The PSS was designed to evaluate patients' attitudes towards nurses and nursing. It is a 25 items Likert- type summated rating scale with three dimensions of patient satisfaction: technical- professional care, educational relationship, and trusting relationship. Both positive and negative items were included in each subscale. Each question was assessed on a five-point Likert measurement scale ranging from "Strongly agree" (=5) to "Strongly disagree" (=1). The higher the PSS score is, the higher is the patient satisfaction with the nursing care provided (Hinshaw and Atwood 1982).

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Nursing / Department of Adult Health Care, Irbid, Jordan

IPD SHARING:
Plan to Share IPD: No
not planned yet